CLINICAL TRIAL: NCT06921811
Title: Bioavailability of Macronutrients and Bioactive Compounds From Chickpea Meals: an Ileostomy Study.
Brief Title: Bioavailability From Chickpea Meals in Ileostomists?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: REC/24/0083
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Nutrition; Absorption; Polyphenolic Compounds and Metabolism; Polyphenols Absorption Profile; Energy Availability
Keywords: Food structure; Cell walls; Macronutrients; Chickpeas; Bioactive compounds

STUDY DESIGN:
Intervention Model Description: Randomised single-blind crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTACT meal (Experimental)
  Interventions: Other: Intact chickpeas
- BROKEN meal (Experimental)
  Interventions: Other: Broken chickpeas

INTERVENTIONS:
Other: Intact chickpeas — Salad meal containing intact chickpeas
  Arms: INTACT meal
Other: Broken chickpeas — Burger meal containing chickpea flour
  Arms: BROKEN meal

SUMMARY:
The matrix of a food can significantly affect how well humans can absorb and use nutrients. Plants like fruits, vegetables, nuts, grains, and legumes have cell walls that form a network around their cells. These cell walls are a barrier for the digestive system to break down completely, which can make it harder to digest the food and get energy from it. This study will explore how the integrity of plant cell walls affects how well humans can absorb macronutrients (protein, fat and carbohydrates) and beneficial compounds e.g. phytochemicals. The study will compare two chickpea meals that have similar nutrients and energy content but differ in the amount of intact plant cell walls e.g. chickpea salad meal (INTACT diet) and chickpea burger meal (BROKEN diet).

DETAILED DESCRIPTION:
The energy content of food can be in principle calculated by multiplying the content of each energy-yielding substrate by the corresponding heat of combustion. However, only part of this energy yielding substrates is converted to energy because of their incomplete digestion and absorption in the gastrointestinal tract. The structural composition of foods, known as the food matrix, significantly affects nutrient bioavailability. One such structural feature is the integrity of plant tissues characterised by the interconnected, continuous network of cell walls which surround and protect plant cells. When cellular integrity is retained, macronutrients are naturally "encapsulated" within cell walls which effectively reduces the rate and the extent of their digestibility by 6-7% compared to a diet poor in plant-based foods. This study aims to investigate the effect of plant tissue integrity on the total energy excretion of a diet, bioavailability of macronutrients and bioactive compounds, and on plasma levels of glucose, essential amino acids and triglycerides. The investigators will do this by comparing two diets which have (approximately) the same composition in macronutrients and energy but different levels of plant tissues integrity, namely a diet rich in intact plant tissues (INTACT diet), and a diet poor in such intact plant tissues (BROKEN diet). The investigators will use an ileostomy model to be able to determine the difference in energy excretion at the level of the terminal ileum.

ELIGIBILITY:
Inclusion Criteria:

* Previously had an ileostomy
* ≥1.5-years post-operative
* Aged 18-60 years
* Males and females (not currently pregnant/lactating)
* Non-smokers
* Not allergic to nuts and celery

Exclusion Criteria:

* Never had an ileostomy
* <1.5-year post-operative
* Not aged 18-60 years
* Pregnant/lactating female
* Smokers
* Allergic to nuts and celery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Ileal fluid energy content | Change over 8 hours comparison between treatments
  Energy content calculated by dry matter (g/100g dry basis)

SECONDARY OUTCOMES:
Ileal fluid macronutrient content | Change over 8 hours comparison between treatments
  Measured by dry matter (g/100g dry basis)
Ileal fluid alkylresorcinol content | Change over 8 hours comparison between treatments
  Measured by Mass Spec
Ileal fluid carotenoid content | Change over 8 hours comparison between treatments
  Measured by Mass Spec
Circulating glucose concentration | Change over 8 hours comparison between treatments
  Blood concentrations of glucose using glucometer
Urinary phenolic content | Change over 8 hours comparison between treatments
  Phenolic concentration e.g. hippuric acid in urine
Circulating insulin, levels | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating essential amino acid levels | Change over 8 hours comparison between treatments
  Blood concentrations of amino acids
Circulating triglyceride levels | Change over 8 hours comparison between treatments
Circulating levels of GLP-1 | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating levels of GIP | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating levels of ghrelin | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating levels of CKK | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating levels of leptin | Change over 8 hours comparison between treatments
  Measured by ELISA in μg/mL.
Circulating levels of bioactive peptides | Change over 8 hours comparison between treatments
  Blood concentrations of legume bioactives

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, N.Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No